CLINICAL TRIAL: NCT04077749
Title: A Randomized Double Blinded Study of Probiotic Bladder Instillation for Prevention of Catheter Associated UTIs in Chronically Catheterized Patients
Brief Title: Probiotic Bladder Instillation for Prevention of Catheter Associated UTIs in Chronically Catheterized Patients
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The study never started. It was withdrawn from the IRB.
Sponsor: Lahey Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2017-041
Record Dates: First submitted 2019-08-28; First posted 2019-09-04 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental)
  Interventions: Biological: Femdophilus probiotic
- Placebo (Placebo Comparator)
  Interventions: Other: Normal Saline

INTERVENTIONS:
Biological: Femdophilus probiotic — Lactobacillus rhamnosus (GR-1®) and reuteri (RC-14®) species, which is offered as an over the counter probiotic capsule sold under the brand name of Femdophilus dissolved in 50 mL normal saline at room temperature.
  Arms: Probiotic
Other: Normal Saline — 50 mL normal saline at room temperature
  Arms: Placebo

SUMMARY:
The proposed study is a randomized, placebo-controlled clinical trial to test the efficacy of an oral Lactobacillus product dissolved in sterile saline and instilled into the urinary bladder in an attempt to colonize the urinary bladder as well as prevent UTIs.

DETAILED DESCRIPTION:
Patients who use a chronic indwelling urinary catheter to drain their bladder will be randomized to receive intravesical instillations of a Lactobacillus solution or sterile saline at the time of a scheduled monthly catheter exchange. Bacterial colonization and frequency of urinary tract infections will be compared between the two groups.

The Lactobacillus solution will be derived from the combination of Lactobacillus rhamnosus (GR-1®) and reuteri (RC-14®) species, which is offered as an over the counter probiotic capsule sold under the brand name of Femdophilus and manufactured by CHR-Hansen of Denmark (phone: +45 45747474; email: info@chr-hansen.com). The contents of the capsules will be dissolved in 50 mL of normal saline at room temperature within one hour prior to administration and left indwelling in the patient's urinary bladder for 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Chronic indwelling urethral catheter or supra-pubic tube for >6 months
3. Prior symptomatic UTI while catheter in place

Exclusion Criteria:

1. Immunosuppressed (HIV, transplant immunosuppression, uncontrolled diabetes)
2. Active infection (may be considered after treatment of active infection)
3. Prior urosepsis requiring ICU admission
4. Significant gross hematuria resulting from catheter exchanges
5. Supravesical urinary diversion
6. Upper urinary tract anatomical abnormality
7. Obstructing urolithiasis
8. Ongoing antibiotic therapy for non-urological infection
9. Indwelling nephrostomy tube or ureteral stent
10. Radiation cystitis
11. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
Bladder colonization with Lactobacillus | 6 months
  Percent of patients with urine cultures positive for lactobacilli species after 6 months.

IPD SHARING:
Plan to Share IPD: No